CLINICAL TRIAL: NCT03573206
Title: Multi-center, Single Arm Continued Access Protocol to Evaluate the Mid-Bore Venous VCS for the Management of the Femoral Venotomy After Catheter-based Interventions Via 6-12F Procedural Sheaths With Single or Multiple Access Sites Per Limb
Brief Title: AMBULATE Continued Access Protocol to Evaluate the Cardiva Mid-Bore Venous Vascular Closure System (VVCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiva Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTL-0543
Record Dates: First submitted 2018-06-14; First posted 2018-06-29 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Surgical Wound
Keywords: vessel closure; venous access site; femoral venotomy; medium bore; multiple access sites
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: All subjects will receive the study device for femoral venotomy closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Cardiva Medical Mid-Bore VVCS for venous femoral access site closure
  Interventions: Device: Cardiva Mid-Bore Venous Vascular Closure Device (VVCS)

INTERVENTIONS:
Device: Cardiva Mid-Bore Venous Vascular Closure Device (VVCS) — The device will be used to close all femoral venous access sites at the end of the case.

SUMMARY:
The objective of the trial is to demonstrate the safety and effectiveness of the Cardiva Mid-Bore Venous Vascular Closure System (VVCS) in sealing femoral venous access sites at the completion of catheter-based procedures performed through 6-12 Fr introducer sheath, while allowing for one or more of the following: elimination of the Foley catheter, elimination of protamine, or allowing same (calendar) day discharge for the appropriate patient population.

DETAILED DESCRIPTION:
A prospective multi-center, single arm continued access clinical protocol enrolling subjects with multiple femoral venous access sites. All femoral venous access sites will be closed using the Cardiva Mid-Bore VVCS. Subjects will be prospectively evaluated for eligibility in the three study groups in order to answer specific research questions related to safety and effectiveness of the device as it relates to the use of peri-procedural urinary catheters, protamine for reversal of heparin, and same calendar day discharge in a select group of procedure types.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

* Acceptable candidate for an elective, non-emergent catheter-based procedure via the common femoral vein(s) using a 6 to 12 Fr inner diameter introducer sheath
* Must be eligible for at least one of the study groups:

  1. No Urinary Catheter: Candidate to undergo the procedure and bedrest without a urinary catheter
  2. No Protamine: Candidate to receive procedural heparin for anti-coagulation management.
  3. Same Calendar Day Discharge: Expected to undergo a procedure for Supraventricular Tachycardia, Atrial Flutter, Atrial Fibrillation or Ventricular Tachycardia; if heparin is planned, it must be reversed with protamine; and physician is expected to be on site for discharge evaluation

Pre-Operative Exclusion Criteria:

Subjects will be excluded from participating in this study if they meet any of the following criteria prior to initiation of the index procedure:

1. Advanced refusal of blood transfusion, if it should become necessary;
2. Active systemic infection, or cutaneous infection or inflammation in the vicinity of the groin;
3. Pre-existing immunodeficiency disorder and/or chronic use of high dose systemic steroids;
4. Known history of bleeding diathesis, coagulopathy, hypercoagulability, or current platelet count < 100,000 cells/mm3;
5. Severe co-existing morbidities, with a life expectancy of less than 12 months;
6. Currently involved in any other investigational clinical trial that may interfere with the outcomes of this study in the opinion of investigator;
7. Femoral arteriotomy in either limb with any of the following conditions:

   1. access within < 10 days
   2. any residual hematoma, significant bruising, or known associated vascular complications
   3. use of a vascular closure device within the previous 30 days;
8. Femoral venotomy in either limb with any of the following conditions:

   1. access within < 10 days
   2. any residual hematoma, significant bruising, or known associated vascular complications c use of a vascular closure device
9. Any planned procedure involving femoral arterial or venous access in either limb within the next 30 days;
10. Any history of deep vein thrombosis, pulmonary embolism or thrombophlebitis;
11. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
12. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or who are lactating;
13. Extreme morbid obesity (BMI greater than 45 kg/m2) or underweight (BMI less than 20 kg/m2);
14. Unable to routinely walk at least 20 feet without assistance;
15. Known allergy/adverse reaction to bovine derivatives;
16. Administration of low molecular weight heparin (LMWH) within 8 hours before or after the procedure;
17. Planned procedures or concomitant condition(s) that may extend ambulation attempts beyond 2-3 hours, and/or hospitalization time (e.g., staged procedure, serious co-morbidity), in the opinion of the Investigator.

Intra-Operative Inclusion Criteria:

The subject must be eligible for at least one of the following study groups:

1. Same Calendar Day Discharge (all criteria apply):

   * In the Investigator's opinion, the subject is a candidate for Same Calendar Day Discharge per protocol.
   * If procedural heparin is used, it must be reversed at or before venous closure.
   * Physician must be on site for discharge evaluation.
   * Supraventricular Tachycardia (SVT) or Atrial Flutter Subjects: No Additional Criteria
   * Atrial Fibrillation or Ventricular Tachycardia Procedure Subjects: CHADS2 Score is ≤1, as assessed pre-operatively.

     * The subject is not enrolled in the No Protamine Group.
2. No Urinary Catheter:

   • The subject does not have a urinary catheter inserted/indwelling at the end of the procedure, just prior to enrollment.
3. No Protamine:

   * The subject received procedural heparin for anti-coagulation management and did not/will not receive protamine.
   * The subject is not enrolled in the Same Calendar Day Discharge Group

Intra-Operative Exclusion Criteria:

Subjects will be excluded from participating in this study if any of the following exclusion criteria occur during the index procedure:

1. Any attempt at femoral arterial access during the procedure;
2. Any procedural complications that may extend routine recovery, ambulation and discharge times;
3. If the physician deems that a different method should be used to achieve hemostasis of the venous access sites, or that the subject should not attempt ambulation according to the protocol requirements;
4. All venous access sites may must comply with the following exclusion criteria, assessed immediately prior to enrollment:

   1. Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure (e.g., multiple stick attempts, accidental arterial stick with hematoma, "back wall stick", etc.) in any of the study veins;
   2. A procedural sheath < 6 Fr or > 12 Fr in inner diameter is present at time of closure;
   3. A procedural sheath > 12 Fr inner diameter at any time during the procedure.
   4. Venous access site location is noted to be "high", above the inguinal ligament (cephalad to lower half of the femoral head or the inferior epigastric vein origin from the external iliac vein);
   5. Intra-procedural bleeding around sheath, or suspected intraluminal thrombus, hematoma, pseudoaneurysm, or AV fistula;
   6. Length of the tissue tract, the distance between the anterior venous wall and skin, is estimated to be less than 2.5 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin M Al-Ahmad, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (3):
- United States (3):
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Valley Hospital, Ridgewood, New Jersey
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 168
Completed | 168
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 164
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 158
  More than one race | 0
  Unknown or Not Reported | 5
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Procedure Success - Effectiveness
Description: Final hemostasis at all venous access sites and freedom from major venous access site closure-related complications through 30 days follow-up
Time Frame: 30 (+/- 10) days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 168
Participants | 168

2. Primary Outcome: Major Venous Access Site Closure-related Complications - Safety, Number of Limbs With Each Event
Description: Rate of combined major venous access site closure-related complications. The method used to determine what would be considered "major" venous access site closure-related complications are those complications which were attributed directly to the closure method used for the access site at the end of the procedure.
Time Frame: 30 (+/- 10) days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 168
Participants | 0

3. Secondary Outcome: Study Group Success Rate - No Urinary Catheter Group, Number of Participants
Description: No peri-procedural urinary catheter insertion required through successful Ambulation (per-patient analyses)
Time Frame: From start of procedure through successful ambulation, assessed to be within 6 hours of final hemostasis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 165
Participants | 161

4. Secondary Outcome: Study Group Success Rate - No Protamine Group, Number of Participants
Description: No delay in Ambulation due to access site bleeding in subjects who receive heparin but are not reversed with protamine (per-patient analyses)
Time Frame: From time of final hemostasis through successful ambulation, assessed to be within 6 hours of final hemostasis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 41
Participants | 39

5. Secondary Outcome: Study Group Success Rate - Same Calendar Day Discharge Group, Number of Participants
Description: Discharge within the same calendar day from the start of the procedure without the need for re-hospitalization within 72 hours of hospital discharge due to access site complications (per-patient analyses)
Time Frame: Within 72 hours post-discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 18
Participants | 18

6. Secondary Outcome: Number of Devices With Success
Description: The ability to deploy the delivery system, deliver the collagen, and achieve hemostasis with the Mid-Bore VVCS (per-access site analyses)
Time Frame: Evaluated for each access site immediately after device delivery is attempted, reported within 5 minutes of deployment
Measure: Count of Units; unit: devices
Units Other Than Participants: devices
Arm/Group | Treatment Arm
Number analyzed (Participants) | 168
Number analyzed (devices) | 622
devices | 612

7. Secondary Outcome: Minor Venous Access Site Closure-related Complications, Number of Limbs With Each Event
Description: Rate of combined minor venous access site closure-related complications. The method used to determine what would be considered "minor" venous access site closure-related complications are those complications which were attributed directly to the closure method used for the access site at the end of the procedure.
Time Frame: 30 (+/- 10) days post-procedure
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | Treatment Arm
Number analyzed (Participants) | 168
Number analyzed (limbs) | 325
limbs | 318

ADVERSE EVENTS:
Time Frame: 30 days (± 10 days)
Description: Access-site related adverse events included
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/168
Serious Adverse Events (participants affected / at risk) | 3/168
Other Adverse Events (participants affected / at risk) | 9/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=168)
Access site closure-related serious adverse events, excluding major and minor complications (Blood and lymphatic system disorders) | 1 (1) — Access site venous re-bleeding after initial hemostasis confirmed for 5 minutes
Access site closure-related serious adverse events, including minor complications (Blood and lymphatic system disorders) | 1 (1) — Access site-related hematoma > 6 cm documented by ultrasound
Access site closure-related serious adverse events, including minor complications (Cardiac disorders) | 1 (1) — Pseudoaneurysm requiring thrombin/fibrin adhesive injection or ultrasound-guided compression
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=168)
Access site venous re-bleeding after initial hemostasis confirmed for 5 minutes (Blood and lymphatic system disorders) | 4 (7) — Access site venous re-bleeding after initial hemostasis confirmed for 5 minutes
Access site-related tissue tract oozing - prolonged* (Surgical and medical procedures) | 1 (1) — Access site-related tissue tract oozing - prolonged*
Access site hematoma ≤ 6 cm (Blood and lymphatic system disorders) | 3 (3) — Access site hematoma ≤ 6 cm
Bruising at the access site* (Surgical and medical procedures) | 1 (1) — Bruising at the access site*
Pain at the access site (Surgical and medical procedures) | 1 (1) — Pain at the access site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03573206/Prot_SAP_ICF_000.pdf